CLINICAL TRIAL: NCT03587350
Title: A Single Site, Pilot Study to Assess the Efficacy of a Novel Minimally Invasive Device to Monitor Dystonic Movements in Patients With Cervical Dystonia Receiving Botulinum Toxin Therapy
Brief Title: Assessing Cervical Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NE16/88973
Record Dates: First submitted 2018-06-28; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Treatment (Active Comparator)
  Interventions: Device: Shimmer monitoring
- Usual care (No Intervention)

INTERVENTIONS:
Device: Shimmer monitoring — The shimmer monitor, monitors movement and the range of movement.
  Arms: Interventional Treatment

SUMMARY:
The study involves the use of a novel, non-invasive, monitoring device to measure the response to treatment with botulinum toxin injections in 24 (16 Intervention and 8 control) patients with cervical dystonia. A baseline assessment, prior to botulinum treatment,will be structured around validated clinical rating scales for cervical dystonia and questionnaires and the performance of simple neck movements, and will be undertaken while the patient wears a movement sensor attached to the head with an elastic strap. The same assessments will be undertaken at 0, 3, 6, 9 and 12 weeks following treatment to assess response. The patients' treatment will not be affected by their participation in the research. The device readings will then be compared with the clinical ratings to establish whether it might be used as a more sensitive measure of treatment response than clinical assessment alone. This will help clinicians to plan and execute botulinum injections more effectively in future

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 years or older (no upper age limit) and willing and able to provide informed consent.
* Participant is able and willing to comply with the follow-up schedule and protocol.
* Participants diagnosed with cervical dystonia.
* Participant has previously received botulinum toxin therapy for cervical dystonia without adverse side effects OR is naïve to botulinum toxin therapy but is suitable to participate in the investigator's opinion

Exclusion Criteria:

* -Participated in another clinical investigation within 30 days.
* Allergy to device components or botulinum toxin.
* Medical co-morbidities that preclude botulinum toxin therapy.
* Patient is incapable of understanding or responding to the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Successful monitoring of movement by the shimmer monitor | 3, 6, 9 and 12 weeks post botulinum therapy
  Accurate assessment of cervical dystonia at different time points to assess change over allocated time frame.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom